CLINICAL TRIAL: NCT01464268
Title: Transepithelial Corneal Collagen Crosslinking for Keratoconus and Corneal Ectasia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cornea and Laser Eye Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLEI-EpiCXL
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Keratoconus; Corneal Ectasia
Keywords: Keratoconus; Corneal Ectasia; Collagen Crosslinking; Riboflavin
MeSH Terms: conditions — Keratoconus | interventions — Riboflavin; Dextrans

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Riboflavin drops every minute (Active Comparator): Administration of riboflavin every 2 minutes for the duration of UV exposure.
  Interventions: Drug: Riboflavin
- Riboflavin drops every 2 minutes (Active Comparator): Administration of riboflavin every 1 minute for the duration of UV exposure.
  Interventions: Drug: Riboflavin

INTERVENTIONS:
Drug: Riboflavin — Administration of riboflavin every 2 minutes for the duration of UV exposure.
  Other Names: Riboflavin without dextran
  Arms: Riboflavin drops every 2 minutes
Drug: Riboflavin — Administration of riboflavin every 1 minute for the duration of UV exposure.
  Other Names: Riboflavin without Dextran
  Arms: Riboflavin drops every minute

SUMMARY:
Corneal collagen crosslinking (CXL) has been proposed as an effective method of reducing progression of both keratoconus and corneal ectasia after surgery, as well as possibly decreasing the steepness of the cornea in these pathologies. During previous studies of the CXL procedure, the surface epithelial cells have been removed. Transepithelial crosslinking in which the epithelium is not removed has been proposed to offer a number of advantages over traditional crosslinking including an increased safety profile by reducing the risk for infection as no epithelial barrier will be broken, faster visual recovery and improved patient comfort in the early postoperative healing period.

DETAILED DESCRIPTION:
The objective of this study is to investigate the difference between two regimens of transepithelial crosslinking. The study will compare two riboflavin dosing regimens during the crosslinking procedure. The primary objective of this study is to evaluate the safety and efficacy of transepithelial corneal collagen crosslinking performed with riboflavin 0.1% for reducing corneal curvature. Safety and efficacy outcomes will then be compared between the treatment groups. In particular, we will compare the two groups with regard to their efficacy in reducing corneal curvature. Secondary outcomes will include visual acuity. Safety assessments will include a tabulation of adverse events, patient symptoms, loss of visual acuity, changes in endothelial cell density, slit lamp examination of the cornea and lens, and contact lens tolerance for contact lens wearers

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* A diagnosis of keratoconus or a diagnosis of corneal ectasia after corneal refractive surgery
* Vision with contact lenses or glasses is worse than 20/20
* Corneal thickness greater than 375 microns at the thinnest point

Exclusion Criteria:

* Eyes classified as either normal, atypical normal, or keratoconus suspect on the severity grading scheme.
* Corneal pachymetry ≤ 350 microns at the thinnest point measured by Pentacam in the eye(s) to be treated.
* Previous ocular condition (other than refractive error) in the eye(s) to be treated that may predispose the eye for future complications
* Clinically significant corneal scarring in the CXL treatment zone
* Pregnancy (including plan to become pregnant) or lactation during the course of the study
* A known sensitivity to study medications
* Patients with nystagmus or any other condition that would prevent a steady gaze during the CXL treatment or other diagnostic tests.
* Patients with a current condition that, in the investigator's opinion, would interfere with or prolong epithelial healing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2011-11; Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Keratometry | 12 months
  The change in maximum keratometry (Kmax) from baseline will be evaluated at 12 months for all eyes randomized to the two treatment groups. As a secondary analysis of this endpoint, the change in maximum keratometry (Kmax) from baseline will be evaluated at 1, 3 and 6 month for all eyes

SECONDARY OUTCOMES:
Manifest refraction | 12 months
  The change in manifest refraction spherical equivalent from baseline will be evaluated at 12 months. As a secondary analysis of this endpoint, a repeated measures analysis of variance will be conducted to assess the profile of the treatments across time at 1,3, and 6 months to look at the effect of wound healing on this variable.
Visual Acuity | 12 months
  Change in BSCVA (best spectacle corrected visual acuity) and UCVA (uncorrected visual acuity) compared to the baseline examination will be evaluated at 12 months postoperatively. As a secondary analysis of this endpoint, data across time from 1, 3, and 6 months following the CXL procedure will be analyzed.
Endothelial cell density | 12 months
  Endothelial cell count will be obtained using specular microscopy (Konan Medical) prior to CXL treatment and at 12 months postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hersh, MD, Principal Investigator — Cornea and Laser Eye Institute
Locations (1):
- Cornea and Laser Eye Institute, Teaneck, New Jersey, United States

REFERENCES:
- [Background] Hersh PS, Greenstein SA, Fry KL. Corneal collagen crosslinking for keratoconus and corneal ectasia: One-year results. J Cataract Refract Surg. 2011 Jan;37(1):149-60. doi: 10.1016/j.jcrs.2010.07.030. PMID 21183110
- [Derived] Davis SA, Bovelle R, Han G, Kwagyan J. Corneal collagen cross-linking for bacterial infectious keratitis. Cochrane Database Syst Rev. 2020 Jun 17;6(6):CD013001. doi: 10.1002/14651858.CD013001.pub2. PMID 32557558